CLINICAL TRIAL: NCT02015845
Title: Evaluation of Accuvein in Obese Patients
Acronym: AVO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recrutment difficulties
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/19; 2013-A00777-38 (Other: ANSM)
Record Dates: First submitted 2013-12-05; First posted 2013-12-19 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Primary Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Accuvein (Experimental): Use of Accuvein to facilitate placement of peripheral intravenous catheters in obese patients
  Interventions: Device: Accuvein
- Routine technique (Active Comparator): Routine technique used to insert a peripheral intravenous catheters in obese patients.
  Interventions: Device: Routine technique

INTERVENTIONS:
Device: Accuvein
  Arms: Accuvein
Device: Routine technique — Placement of peripheral intravenous catheters using the routine technique
  Arms: Routine technique

SUMMARY:
The objective of this study is to evaluate the effectiveness of Accuvein to facilitate placement of peripheral intravenous catheters in obese patients. This clinical protocol is designed to determine whether using Accuvein increases the ease and efficiency of venous cannulation (as perceived by the operator), decreases the time to effective cannulation, and decreases the patient's perception of the pain.

ELIGIBILITY:
Inclusion Criteria:

* obese adults ( BMI equal or greater 35) requiring a venous blood sampling or the placement of a venous peripheral catheter

Exclusion Criteria:

* pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-11; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Percentage of success of the first vein puncture | one hour
  Successful successful placement of IV catheter

SECONDARY OUTCOMES:
Score of evaluation of the device | one hour
  Evaluation of the device by the operator and the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Hospitalier Franco-Britannique, Levallois-Perret, Hauts de Seine, France